CLINICAL TRIAL: NCT05599516
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial to Evaluate Efficacy, Safety and Immunogenicity of LIBP Recombinant COVID-19 Vaccine (CHO Cell, NVSI-06-09) and BIBP Recombinant COVID-19 Vaccine (CHO Cell, NVSI-06-09) in Healthy Population Aged 18 and Above
Brief Title: Recombinant COVID-19 Vaccine (CHO Cell, NVSI-06-09) Phase III Clinical Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: China National Biotec Group Company Limited (Industry); Lanzhou Institute of Biological Products Co., Ltd (Industry); Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CNBG-REC-2022006
Record Dates: First submitted 2022-10-27; First posted 2022-10-31 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Coronavirus Infections
Keywords: COVID-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 LIBP-Rec-Vaccine Group (Experimental): Subject vaccinated with ≥2 doses of inactivated COVID-19 vaccine for ≥6 months
  Interventions: Biological: LIBP-Rec-Vaccine
- Cohort 1 BIBP-Rec-Vaccine Group (Experimental): Subject vaccinated with ≥2 doses of inactivated COVID-19 vaccine for ≥6 months
  Interventions: Biological: BIBP-Rec-Vaccine
- Cohort 1 placebo control group (Placebo Comparator): Subject vaccinated with ≥2 doses of inactivated COVID-19 vaccine for ≥6 months
  Interventions: Biological: placebo
- Cohort 2 LIBP-Rec-Vaccine Group (Experimental): Subject vaccinated with ≥2 doses of mRNA COVID-19 vaccine for ≥6 months
  Interventions: Biological: LIBP-Rec-Vaccine
- Cohort 2 BIBP-Rec-Vaccine Group (Experimental): Subject vaccinated with ≥2 doses of mRNA COVID-19 vaccine for ≥6 months
  Interventions: Biological: BIBP-Rec-Vaccine

INTERVENTIONS:
Biological: LIBP-Rec-Vaccine — Intramuscular injection of LIBP-Rec-Vaccine in the deltoid muscle of the upper arm
  Arms: Cohort 1 LIBP-Rec-Vaccine Group; Cohort 2 LIBP-Rec-Vaccine Group
Biological: BIBP-Rec-Vaccine — Intramuscular injection of BIBP-Rec-Vaccine in the deltoid muscle of the upper arm
  Arms: Cohort 1 BIBP-Rec-Vaccine Group; Cohort 2 BIBP-Rec-Vaccine Group
Biological: placebo — Intramuscular injection of placebo in the deltoid muscle of the upper arm
  Arms: Cohort 1 placebo control group

SUMMARY:
This clinical trial adopts a randomized, double-blind and placebo-controlled design.

A total of 16000 participants are planned to be enrolled, of which, Cohort 1: 15000 participants vaccinated with ≥2 doses of inactivated COVID-19 vaccine for ≥6 months will be randomly administered at ratio of 1:1:1 with 1 dose of LIBP-Rec-Vaccine, BIBP-Rec-Vaccine or placebo intramuscularly to the deltoid muscle of upper arm.

Cohort 2: 1000 participants vaccinated with ≥2 doses of mRNA COVID-19 vaccine for ≥6 months will be randomly administered at ratio of 1:1 with 1 dose of LIBP-Rec-Vaccine or BIBP-Rec-Vaccine intramuscularly to the deltoid muscle of upper arm.

ELIGIBILITY:
Inclusion Criteria:

* Age range: healthy population aged ≥18;
* Judged by the investigator that the health condition is well after inquiry and physical examination;
* Cohort 1: participants vaccinated with ≥2 doses of inactivated COVID-19 vaccines for ≥6 months since the last dose of vaccination; Cohort 2: participants vaccinated with ≥2 doses of mRNA COVID-19 vaccines for ≥6 months since the last dose of vaccination;
* Be able and willing to complete all prescribed study schedules during the whole study period;
* The participant himself/herself is able and willing to understand study procedures, sign the informed consent form voluntarily after informed consent and comply to requirements of the study protocol.

Exclusion Criteria:

* Symptomatic and suspected COVID 19 infection positive ;
* Urine pregnancy test is positive; Women of childbearing age who have positive urine pregnancy test, who are pregnant, lactating, or women who have planned pregnancy within 6 months;
* Auxiliary temperature before vaccination is ≥37.3℃ (tympanic/forehead temperature ≥37.8℃);
* Previous allergy history of vaccine vaccination (such as acute allergic reaction, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain, etc.) or allergy to known components of COVID-19 vaccine;
* Have a history of hospital-diagnosed thrombocytopenia or other coagulation disorders;
* With known immunological impairment or compromised immunological function diagnosed by the hospital;
* Received whole blood, plasma and immunoglobulin therapy within 1 month;
* Known or suspected of suffering from the following diseases: acute or chronic active respiratory diseases, severe cardiovascular diseases [cardiopulmonary failure, hypertension uncontrollable by drugs (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 95 mmHg)], acute infection, active phase of chronic disease, liver and kidney diseases, severe diabetes, malignant tumor, infectious skin diseases or severe skin allergy, HIV infection, etc. (Examination report can be provided)
* Received live attenuated vaccine within one month before vaccination;
* Received inactivated vaccine within 14 days before vaccination;
* Other contraindications related to vaccination that investigators believe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16000 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Efficacy of LIBP-Rec-Vaccine/ BIBP-Rec-Vaccine against COVID-19 of immunization in healthy population aged 18 and above. | 14th day after vaccination
  Rates of cohort 1 subjects not infected with COVID-19

SECONDARY OUTCOMES:
Cohort 1: Efficacy of LIBP-Rec-Vaccine /BIBP-Rec-Vaccine against COVID-19 asymptomatic infection in healthy population aged 18 and above | 14th day after vaccination
  Rates of cohort 1 subjects who are not asymptomatic infection with COVID-19
Cohort 1: Efficacy of LIBP-Rec-Vaccine /BIBP-Rec-Vaccine against COVID-19 severe cases in healthy population aged 18 and above | 14th day after vaccination
  Rates of cohort 1 subjects who are not severe cases with COVID-19
Cohort 1: Efficacy of LIBP-Rec-Vaccine / BIBP-Rec-Vaccine against COVID-19 related deaths in healthy population aged 18 and above. | 14th day after vaccination
  Rates of cohort 1 subjects who are not related deaths with COVID-19
GMT of subject's anti-SARS-CoV-2 neutralizing antibody is non-inferior to that of Cohort 1（ LIBP-Rec-Vaccine / BIBP-Rec-Vaccine） | 14th day after vaccination
  Cohort 2 Immunogenicity subgroup only
GMT of subject's anti- SARS-CoV-2 neutralizing antibody | 14th day、28th day after vaccination
  Immunogenicity subgroup only
GMI of subject's anti- SARS-CoV-2 neutralizing antibody | 14th day、28th day after vaccination
  Immunogenicity subgroup only
4-fold increase rate of subject's anti- SARS-CoV-2 neutralizing antibody | 14th day、28th day after vaccination
  Immunogenicity subgroup only
GMT of subject's anti- SARS-CoV-2 neutralizing antibody | 3th month、6th month after vaccination
  Immunogenicity subgroup only
GMI of subject's anti- SARS-CoV-2 neutralizing antibody | 3th month、6th month after vaccination
  Immunogenicity subgroup only
4-fold increase rate of subject's anti- SARS-CoV-2 neutralizing antibody | 3th month、6th month after vaccination
  Immunogenicity subgroup only
The incidence and severity of any adverse reactions | within 30 minutes after vaccination
The incidence and severity of solicited adverse events | within 30 minutes after vaccination
The incidence and severity of solicited adverse reactions | within 0-7 days after vaccination
The incidence and severity of unsolicited adverse reactions | within 0-7 days after vaccination
The incidence and severity of solicited adverse reactions | within 8-30 days after vaccination
The incidence and severity of solicited adverse events | within 8-30 days after vaccination
The incidence of SAE observed | Within 6 months of vaccination
The incidence of AESI observed | Within 6 months of vaccination
Cross-neutralizing effect of recombinant COVID-19 vaccine against different variants (prototype strain, Delta, Omicron and other potential emerging dominant circulating variants) | 14th day after vaccination
  Immunogenicity subgroup only

OTHER OUTCOMES:
Subject's the genotypes of SARS-CoV-2 virus in endpoint cases | During the study, approximately 14 months
Explore the occurrence of ADE/VED following immunization with LIBP-Rec-Vaccine and BIBP-Rec-Vaccine | During the study, approximately 14 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Khalifa Medical City, SEHA, Abu Dhab, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No